CLINICAL TRIAL: NCT02418039
Title: Effect of a High Protein Diet Versus Normal Protein Diet in Treating Patients With Minimal Hepatic Encephalopathy. Double-blind Clinical Trial
Brief Title: High Protein Diet Versus Normal Protein Diet in Treating Patients With Minimal Hepatic Encephalopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of the reconversion of the hospital to care for patients with COVID19. For this reason, it was not possible to continue recruiting and monitoring patients for this clinical study.
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Segundo Moran Villota, Asociado B, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2014-785-007
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Liver Cirrhosis
Keywords: Minimal hepatic encephalopathy; Nutrition
MeSH Terms: conditions — Liver Cirrhosis | interventions — Diet, High-Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MHE and normal protein diet (Placebo Comparator): Normal protein content (0.8 g/kg/day)
  Interventions: Dietary Supplement: Normal protein
- MHE and high protein diet (Experimental): Patients with minimal hepatic encephalopathy will received a high protein diet (1.5 g/kg/day)
  Interventions: Dietary Supplement: High protein diet

INTERVENTIONS:
Dietary Supplement: High protein diet — It has been suggested that administrating a high protein diet in patients with liver cirrhosis and with minimal hepatic encephalopathy could prevent the development of malnutrition, increase the detoxification of ammonia by the muscle to consequently delay the onset overt hepatic encephalopathy and prolong patient survival. However, information is scarce and inconclusive regarding the potential role of dietary protein in the prevention and treatment of minimal hepatic encephalopathy.
  Other Names: hyperproteic diet
  Arms: MHE and high protein diet
Dietary Supplement: Normal protein — A normal protein diet will be administrated in patients with MHE.
  Arms: MHE and normal protein diet

SUMMARY:
A total of 80 patients diagnosed with liver cirrhosis and minimal hepatic encephalopathy will be recruited. They will be randomized to receive high protein diet ( n = 40) and a normal protein diet ( n = 40 ) during one month. Randomization will be conducted by an external monitor and will keep the secret codes until the end of the study. All patients will be provided with structured menus and two snacks a day as an amaranth protein supplement. The supplement will content the same amount of fiber but the protein content will vary depending on the group to which the patient is assigned.

DETAILED DESCRIPTION:
The protein in the diet is a major source of ammonia in blood, which is considered one of the factors involved in the pathogenesis of hepatic encephalopathy. However ; it is also known than the restriction on the consumption of protein predisposes to depletion of muscle mass, and increase the risk to develop overt hepatic encephalopathy, due to the muscle role in the detoxification of ammonia in presence of liver failure. Currently, the type and amount of protein in the diet to treat minimal hepatic encephalopathy (MHE) is unknown. In this study, the investigators will administrated two types of protein content in patients with MHE: a high protein diet (1.5 g/kg/day) vs a normal protein diet (0.8 g/kg/day) during 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis of any etiology
* Men and women between 18 and 70 years.
* Right-holders of the Mexican Social Security Institute
* Patients who agree to participate in the study and signed the informed consent

Exclusion Criteria:

* Recent history of alcohol abuse and/or drugs (less than 6 weeks).
* Illiterate
* Alcoholic cirrhosis
* History and/or diagnosis of overt hepatic encephalopathy
* Consumption of psychotropic medications (benzodiazepines, antiepileptics)
* Patients under treatment with lactulose, lacitol, rifaximin, neomycin, metronidazole and/or fiber supplements.
* History of chronic renal disease or heart failure
* Patients with gastrointestinal bleeding
* History of neurological or psychiatric disorders that affect the ability to develop neuropsychological tests
* Diagnosis of bacterial overgrowth
* Diagnosis of liver cancer
* Patients with ophthalmologic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Reversal of minimal hepatic encephalopathy intervention) | 1 month
  Number of patients who reverts the minimal hepatic encephalopathy after dietary intervention

SECONDARY OUTCOMES:
Nutritional Status | 1 month
  To evaluate the effect of dietary intervention on nutritional status. The nutritional status will be evaluated with the hand strength measured by a dynamometer. A value less than 30 kg will be consider as risk of malnutrition.
Incidence of hepatic encephalopathy | 1 month
  Number of patients that develop minimal hepatic encephalopathy after dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Segundo Moran, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico